CLINICAL TRIAL: NCT02879357
Title: Palliative Care Population Management Project for Integrated Care Management Program for High-Risk Patients
Acronym: iCMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners HealthCare (Other)
Responsible Party: Principal Investigator, Bernacki, Rachelle E.,M.D., Rachelle Bernacki, M.D., M.S., Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P000211
Record Dates: First submitted 2015-05-07; First posted 2016-08-25 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Failure to Thrive
Keywords: Care management; end of life; advanced care planning; palliative care
MeSH Terms: conditions — Failure to Thrive; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trained Clinicians (Experimental): Training in Serious Illness Communication Guide
  Interventions: Behavioral: Training
- Untrained Clinicians (No Intervention): No training in Serious Illness Communication Guide

INTERVENTIONS:
Behavioral: Training — 1. Clinician training
  2. System for patient selection
  3. System of "triggering" and tracking conversations
  4. Training on how to use the Serious Illness Care Guide, a guide for patients about initiating conversations with family members about end-of-life goals and values
  5. Longitudinal Medical Record (LMR) documentation module to serve as a "Single source of truth" about advance care preferences in the LMR.
  Arms: Trained Clinicians

SUMMARY:
The hypothesis of the Serious Illness Care Program (SICP) is that adherence to the Serious Illness Conversation Guide (SICG) portion, the SIGC, will enhance patient understanding and allow control over their own decisions, relieve burdens of decision-making on family members, and help patients achieve a state of peace as they approach the end of life.

DETAILED DESCRIPTION:
The aim of the Serious Illness Care Program (SICP) is to provide clinicians with an evidence-based structure for eliciting and documenting vital information about preferences for patient driven care of their serious illness. It is designed to help open the door for patients, families, and clinicians to talk and reflect on end-of-life issues in an ongoing way. The hypothesis of the Serious Illness Care Program is that adherence to the conversation guide portion, the SIGC, will enhance patient understanding and allow control over their own decisions, relieve burdens of decision-making on family members, and help patients achieve a state of peace as they approach the end of life. For this protocol specifically, the investigators are testing a pilot intervention of a quality improvement project; the investigators plan to train clinicians and assess the feasibility and impact of the Serious Illness Care Program, which includes patient identification, clinician training, "triggering" of clinicians to conduct the SICG conversation, and documentation, in the iCMP at the Brigham and Women's Hospital.

ELIGIBILITY:
Clinician Inclusion Criteria:

1. Brigham and Women's Hospital or Newton Wellesley Primary Care Clinician at one of the following practices: The Phyllis Jen Center for Primary Care, Faulkner Community Physicians, Brigham and Women's Physician Group, Brigham & Women's Primary Care Associates of Brookline, Brigham Circle Medical Associates, Faulkner
2. Care for patients enrolled in Brigham and Women's Hospital integrated Care Management Program (iCMP)

Clinician Exclusion Criteria:

1. Resident in Training
2. Non-English Speaking Clinic (e.g. Spanish Clinic)

Patient Inclusion Criteria:

1. Over 18 years of age
2. English Speaker
3. Patient at Brigham and Women's Hospital or Newton Wellesley Primary Care Clinician at one of the following practices: The Phyllis Jen Center for Primary Care, Faulkner Community Physicians, Brigham and Women's Physician Group, Brigham & Women's Primary Care Associates of Brookline, Brigham Circle Medical Associates, Faulkner
4. Enrolled in Brigham and Women's Hospital integrated Care Management Program

Patient Exclusion Criteria:

1. Patient at Dana-Farber Cancer Institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible patients with documented goals of care conversations | from date of determination of eligibility to date of death death during the study period, assessed for up to 18 months
  For patients whose death falls during the study period, the percentage of goals of care conversations completed and documented in the electronic medical record by clinicians in the intervention group and the control group. A completed conversation is defined by key elements being documented regarding goals of care in the patient's medical record.

SECONDARY OUTCOMES:
Median number of days before death of first documented goals of care conversation | from date of determination of eligibility to date of death during the study period, assessed for up to 18 months
  For all patients whose death falls during the study period, the median number of days from the date of the first documented goals of care conversation to date of death in both the intervention and the control group.
Percentage of eligible patients with more comprehensive documentation of goals of care before death | from date of determination of eligibility to date of death during study period, assessed for up to 18 months
  For all patients whose death falls during the study period, the percentage of patients with more comprehensive goals of care documentation before death in both the intervention group and the control group. More comprehensive is defined as documentation of a goals of care conversation that addresses more than code status only and will be evaluated for completeness in containing more key elements of a Serious Illness Care Guide conversation.

OTHER OUTCOMES:
Completion of eligible conversations | from date of clinician training study start to study end date, assessed for up to 18 months
  Median percentage of eligible patients with completed conversations (will report for all intervention clinicians as a whole and also on individual clinician level)
Length of conversation | from date of clinician training study start to study end date, assessed for up to 18 months
  Median length of time per conversation in the intervention group as reported by clinician survey
Clinician Confidence | at initial clinician training and end of study (an average of 18 months)
  Clinicians who are trained to use the Guide will have improved confidence in carrying out end-of-life conversations, compared to untrained clinicians. Confidence will be evaluated before training and at end of study and measured using a 22-question survey asking clinicians to quantify their confidence on a scale of 1-7. This survey was designed by study investigators based on national surveys used to evaluate a sample of medical students, residents, and attending physicians' attitudes about end-of-life care, as well as the Harvard Medical School Center for Palliative Care's national faculty development program.
Clinician Attitudes | at clinician training and end of study (an average of 18 months)
  Clinicians who are trained to use the Guide will have improved attitudes in carrying out end-of-life conversations, compared to untrained clinicians. Confidence will be evaluated before training and at end of study and measured using an 11-question survey asking clinicians to quantify their confidence on a scale of 1-5. This survey was designed by study investigators based on national surveys used to evaluate a sample of medical students, residents, and attending physicians' attitudes about end-of-life care, as well as the Harvard Medical School Center for Palliative Care's national faculty development program.
Utilization | at end of study (an average of 18 months)
  Patients of clinicians who are trained to use the Guide will have higher rates of hospice usage, less health care utilization, and lower expenses near the end of life. We will measure utilization outcomes for those patients for whom we have claims data through risk contracts and the accountable care organization and will compare usage and trends between intervention and comparison patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle E Bernacki, MD, Principal Investigator — Dana-Farber Cancer Institute; Susan D Block, MD, Principal Investigator — Dana-Farber Cancer Institute; Rebecca Cunningham, MD, Principal Investigator — Brigham and Women's Hospital; Joshua R Lakin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No